CLINICAL TRIAL: NCT05807568
Title: MIStreatment Screening in Elders Before Discharge (MISSED) Study
Brief Title: MIStreatment Screening in Elders Before Discharge
Acronym: MISSED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julia A Hiner, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-22-1009
Record Dates: First submitted 2023-03-27; First posted 2023-04-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Elder Abuse; Surveys and Questionnaires; Self Neglect; Geriatrics; Geriatric Assessment; Health Services for the Aged; Aged
Keywords: Elder Mistreatment; Abuse; Neglect; Exploitation; Screening; Geriatric; Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCAEM EM-SART Pre-Screen (Experimental)
  Interventions: Other: NCAEM EM-SART Pre-Screen

INTERVENTIONS:
Other: NCAEM EM-SART Pre-Screen — Participants will be verbally asked the 3 participant questions on the NCAEM EM-SART Pre-Screen either directly or with support of hospital approved telephonic interpreters. Answers will be documented by the investigator digitally. Participants will be interviewed one time for a duration of approximately 15 minutes. No further action will be taken on study participants with negative elder mistreatment screens, unless findings concerning for emotional distress are identified by the investigator. If emotional distress is identified, these observations will be communicated to Geriatric Medicine team in person or via secure/encrypted email, with recommendations to follow-up with the participant about the results and take appropriate care actions. Study participants with positive elder mistreatment will have results shared with the study participant directly and with the Geriatric Medicine primary team via secure/encrypted email.

SUMMARY:
The purpose of this study is to demonstrate the feasibility of introducing, implementing, and integrating a brief, existent elder mistreatment screening tool (the National Collaboratory to Address Elder Mistreatment (NCAEM)'s Elder Mistreatment - Screening And Response Tool (EM-SART) Pre-Screen) in the Memorial Herman Hospital (MHH)-Texas Medical Center (TMC)Acute Care of Elders(ACE) (MHH-TMC ACE) unit and to identify older adults who may already be suffering from abuse, neglect, and/or financial exploitation, as well as connecting the study participants to the primary Geriatric Medicine team on the ACE unit such that additional care, evaluation (including additional in-depth mistreatment screening), and intervention can be taken to prevent and minimize further harm prior to discharge. The investigators hope to reduce missed opportunities for mistreatment detection to lead to safer health outcomes and hospital discharges.

ELIGIBILITY:
Inclusion Criteria:

* current admission to the MHH-TMC ACE unit
* ability to independently hear, understand, and verbally answer the 3 participant questions on the NCAEM's EM-SART Pre-Screen screening tool when it is read to them

Exclusion Criteria:

* unwillingness to participate in the research study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Number of units using this NCAEM EM-SART Pre-Screen tool | 12 months after study
  How many times the NCAEM EM-SART Pre-Screen tool is attempted with consented patients
Number of participants who have identified elder mistreatment | 15 minute evaluation of each participant, no follow-up
  Study participants screening positive based on NCAEM EM-SART Pre-Screen tool

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Hiner, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No